CLINICAL TRIAL: NCT05493241
Title: Development and Feasibility of a Behavioral Activation Intervention to Support Independence in Older Veterans at Risk for Functional Decline
Brief Title: Behavioral Activation for Independence in Older Veterans
Acronym: ACTIVaTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3930-W
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Functional Independence
Keywords: functional status; aged; psychosocial intervention; Veterans

STUDY DESIGN:
Intervention Model Description: Participants in Aim 2 (open trial, single arm) will all receive the ACTIVaTE intervention. Participants in Aim 3 (randomized controlled trial) will be randomly assigned to the ACTIVaTE intervention or usual care.
Who Masked: Outcomes Assessor
Masking Description: In Aim 3, a research coordinator masked to group assignment will conduct the 8- and 12-week assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open trial (Other): In Aim 2, all 10 participants will receive the ACTIVaTE intervention.
  Interventions: Behavioral: Behavioral Activation for Independence in Older Veterans (ACTIVaTE)
- ACTIVaTE intervention (Experimental): In Aim 3, 24 participants will be randomized to receive the ACTIVaTE intervention.
  Interventions: Behavioral: Behavioral Activation for Independence in Older Veterans (ACTIVaTE); Other: Usual care
- Usual care (Other): In Aim 3, 24 participants will be randomized to a usual care arm.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Behavioral Activation for Independence in Older Veterans (ACTIVaTE) — 6 sessions delivered by a psychology trainee by telehealth will cover the core content of an existing BA model, Brief Behavioral Activation for Depression-Revised (BATD-R), including education on BA and rationale for the intervention, activity monitoring, values exploration, and activity selection and planning. ACTIVaTE will include the following key modifications: 1) modifying background and psychoeducation to focus on maintaining functional independence; 2) tailoring content to Veterans; 3) adapting materials for VVC telehealth delivery; 4) incorporating elements of activity and environmental modification from an OT perspective; and 5) adding content on VA and community resources for older Veterans. Each session is structured similarly, consisting of education or review of concepts, review of homework and troubleshooting challenges, discussion of core content (e.g. values exploration or activity planning/scheduling), and assignment of homework for the next session.
  Arms: ACTIVaTE intervention; Open trial
Other: Usual care — In this study, both arms will have access to usual care as part of their routine clinical care. Recognizing the heterogeneity of primary care services provided to patients at risk for functional decline, we will minimally standardize the usual care arm by providing a booklet of educational information on maintaining activity to support independence in aging (e.g., an NIH handout "Participating in Activities you Enjoy as you Age" and information on VA and community recreation programs to stay active) that will be mailed to participants after randomization.
  Arms: ACTIVaTE intervention; Usual care

SUMMARY:
As Veterans age, chronic health conditions increase their risk of functional limitations, or difficulty completing day-to-day activities independently. Older adults with functional limitations are more likely to be hospitalized or admitted to long-term care facilities. Maintaining independence at home and in the community is a high priority for many older Veterans. The goal of this study is to support the physical, cognitive, and social functioning of older Veterans by developing a program based on behavioral activation, an evidence-based brief psychosocial intervention that helps individuals increase their engagement in activities aligned with their values (i.e. what matters most to them). The study consists of 3 aims. Aim 1 involves adapting an existing behavioral activation program for older Veterans at risk for functional decline to be delivered by video telehealth and seeking feedback from Veterans and VA staff about the program materials. Aim 2 involves testing the program in a group of 10 Veterans to learn whether it is satisfactory to Veterans; the investigators will make improvements to the program based on the information gathered in this aim. Aim 3 is a randomized controlled trial that will test the behavioral activation program compared to usual care in older adulthood in 48 Veterans. This will help determine whether the program is possible to deliver as planned and acceptable to Veterans, and assess the potential effects of the program on functioning and related health outcomes.

DETAILED DESCRIPTION:
The overarching goal of this study is to develop and test the feasibility and acceptability of a telehealth-delivered behavioral activation (BA) intervention (ACTIVaTE) to promote physical, cognitive, and social functioning in community-dwelling older Veterans at risk for functional decline. This work will provide preliminary data that will inform the design of a future adequately-powered efficacy trial.

This proposal consists of three aims: Aims 1 and 2 are focused on intervention adaptation and refinement of an existing BA model to optimize the acceptability of the ACTIVaTE intervention and study procedures for older Veterans (NIH Stage Model for Behavioral Intervention Development stage IA). Aim 3 is a feasibility pilot RCT of the ACTIVaTE intervention versus usual care (NIH Stage Model stage IB). A focus on Stage I procedures (intervention generation and refinement, including initial feasibility pilot testing) will ensure that the intervention is optimally tailored to the study population and feasible for subsequent stage II-IV efficacy and effectiveness testing. Mixed methods will be used throughout all aims to optimize the intervention for the VA and telehealth delivery, to incorporate Veterans' preference into the intervention and study design, and to understand barriers and facilitators to implementation during the pilot phase.

Aim 1: Adapt BA protocol for ACTIVaTE (Year 1). The investigators will develop ACTIVaTE based on an existing BA model (Behavioral Activation Treatment for Depression-Revised) for delivery to older Veterans at risk for functional decline via the VA's video telehealth platform (VA Video Connect). The previous experience with BA will inform the initial adaptation, incorporating perspectives from primary care, geropsychology, and occupational therapy. The investigators will seek feedback on the preliminary manual and participant workbook via semi-structured interviews with VA psychologists (n=5), occupational therapists (n=5), and Veterans (n=5), using findings from rapid qualitative analysis to further modify the materials. By design, this intervention development aim is hypothesis-generating as opposed to hypothesis-driven, as the investigators will be using qualitative methods to extract themes that will guide intervention adaptation and refine subsequent aims.

Aim 2: Refine the ACTIVaTE intervention (Year 2). Preliminary acceptability of the intervention will be established through a small open trial of the intervention delivered via VVC to 10 older Veterans at risk for functional decline (Vulnerable Elders Survey-13 score 3) recruited from VA primary care. This early acceptability testing will focus on Veteran satisfaction and experience with the intervention and study procedures and will also be used to optimize interventionist training and fidelity assessment. Participants will complete qualitative interviews guided by the Theoretical Framework of Acceptability (TFA) as well as the Client Satisfaction Questionnaire (CSQ) and findings will be used to further refine the intervention materials prior to the pilot RCT. The investigators hypothesize that the intervention will be preliminarily acceptable as determined by high CSQ scores ( 80%) among at least 70% of participants. The investigators also anticipate that themes identified within TFA domains will demonstrate general acceptability with some recommendations to inform refinement.

Aim 3: Determine feasibility, acceptability, and preliminary impact of ACTIVaTE (Years 3-4). The investigators will conduct a 1:1 randomized pilot RCT of ACTIVaTE versus usual care in 48 Veterans at risk for functional decline (VES-13 score 3) recruited from VA primary care. The primary goal of the pilot RCT is to establish feasibility and acceptability, and a fully powered RCT is beyond the scope of this study. However, the investigators will explore preliminary evidence of potential impact on functioning. The investigators will collect clinical measures at baseline, 8 weeks, and 12 weeks, using the Ambulatory Measure for Post-Acute Care (AM-PAC) and PROMIS Satisfaction with Social Roles and Activities as primary measures of physical, cognitive, and social functioning. The investigators will also conduct semi-structured interviews with a purposive sample of participants based on satisfaction and adherence. Exploratory outcomes include objective physical and cognitive function, quality of life, mood, behavioral activation, social isolation, and engagement in physical, cognitive, and social activities.

Aim 3a: Feasibility will be determined by enrollment and retention. Acceptability will be determined by adherence and satisfaction, as well as by themes from qualitative interviews. The investigators hypothesize that the intervention will be feasible (enrollment of 2-3 participants per month for a total n=48; retention of at least 80% of participants at 12 weeks follow-up) and acceptable ( 80% of participants complete at least 5/6 sessions; 70% of participants report high satisfaction on Client Satisfaction Questionnaire).

Aim 3b: Preliminary impact on AM-PAC and PROMIS will be explored through within and between groups mixed-effects linear regression models and proportions of participants who achieve minimal clinically important change in outcomes. The investigators hypothesize that a greater proportion of participants in the ACTIVaTE group will achieve minimal clinically important change in AM-PAC and PROMIS than usual care.

ELIGIBILITY:
Inclusion Criteria:

* Receiving VA primary care
* Community-dwelling (living outside nursing homes)
* At risk for functional decline (VES-13 score 3 or higher); (Aim 3 only) For individuals who are age 85 and score 3 on VES based on age alone, we will also require that they have a score of 0.2 on the VA frailty index (mild frailty or greater)

Exclusion Criteria:

* Non-English speaking
* Currently receiving physical therapy, occupational therapy, or psychotherapy
* Advanced cognitive impairment (MIS-T 3 or lower)
* Uncorrectable hearing or visual impairment that would preclude participation
* Unstable physical or mental health condition:

  * ongoing evaluation of new cardiac or respiratory symptoms
  * receiving hospice or palliative care services
  * anticipated surgery in the next 3 months
  * severe depressive symptoms (PHQ-9 14 or higher)
  * active suicidal ideation
  * likely substance use disorder (positive TICS)
  * schizophrenia
  * psychosis in the past 6 months
* (Aim 2 and 3) Currently receiving physical therapy, occupational therapy, or psychotherapy
* (Aim 3 only) No access to video-capable device (tablet, smartphone, computer) for VVC visits

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Baseline
  Proportion screened who enroll; number or participants enrolled per month; total number of participants enrolled. Enrollment will serve as a measure of feasibility in Aim 3, with a benchmark of 2-3 Veterans enrolled per month to achieve a sample of 48 participants enrolled over 18 months.
Retention at 12 weeks | 12 weeks
  Proportion enrolled who complete 12wk follow-up. Retention will serve as a measure of feasibility in Aim 3, with a benchmark of at least 80% of participants enrolled completing the 12wk follow-up.
Adherence | 12 weeks
  Proportion completing at least 5 of 6 sessions. Adherence will serve as a measure of acceptability in Aim 3 with a benchmark of At least 80% of participants completing 5-6 sessions.
Satisfaction at intervention completion | 6 weeks
  Proportion reporting high satisfaction (at least 80% on the Client Satisfaction Questionnaire [CSQ-8]). Satisfaction at intervention completion (6 weeks) will serve as a measure of acceptability in Aim 2 with a benchmark of at least 70% of participants report high satisfaction. Validated measure of treatment satisfaction in mental health and research settings; raw scores will be transformed to a 100-point percentage scale.
Themes based on Theoretical Framework of Acceptability domains | 6 weeks
  Themes regarding acceptability of the intervention based on the Theoretical Framework of Acceptability as determined by participant semi-structured interviews. This will serve as a measure of acceptability in Aim 2.
Satisfaction at study completion | 12 weeks
  Proportion reporting high satisfaction (at least 80% on the Client Satisfaction Questionnaire [CSQ-8]). Satisfaction at study completion (12 weeks) will serve as a measure of acceptability in Aim 3 with a benchmark of at least 70% of participants report high satisfaction. Validated measure of treatment satisfaction in mental health and research settings; raw scores will be transformed to a 100-point percentage scale.

SECONDARY OUTCOMES:
Recruitment | Baseline
  Proportion approached who agree to screening. Recruitment will serve as a measure of feasibility in Aim 3.
Change in physical functioning as measured by the Ambulatory Measure for Post-Acute Care (AM-PAC) Daily Activities and Basic Mobility Scales | Baseline, 6-8 weeks, 12 weeks
  This standardized measure of physical and cognitive functioning has standardized scores with a mean of 50 and standard deviation of 10; higher scores indicate better functioning. The investigators will measure both change over time and the proportion of participants who achieve clinically meaningful change. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Randomization | Baseline
  Proportion eligible who agree to randomization. Randomization will serve as a measure of feasibility in Aim 3.
Change in cognitive functioning as measured by the Ambulatory Measure for Post-Acute Care (AM-PAC) Applied Cognitive Scale | Baseline, 6-8 weeks, 12 weeks
  This standardized measure of physical and cognitive functioning has standardized scores with a mean of 50 and standard deviation of 10; higher scores indicate better functioning. The investigators will measure both change over time and the proportion of participants who achieve clinically meaningful change. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Fidelity | 12 weeks
  Mean fidelity score on fidelity checklist. Fidelity will serve as a measure of feasibility in Aim 3 with a benchmark of mean fidelity rating at least 80% on intervention checklist.
Change in social functioning as measured by the PROMIS Satisfaction with Social Roles and Activities (Short Form-8a) | Baseline, 6-8 weeks, 12 weeks
  Scores are standardized with a mean of 50 and standard deviation of 10; higher scores indicate better functioning. The investigators will measure both change over time and the proportion of participants who achieve clinically meaningful change. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Barriers and facilitators | 12 weeks
  Themes regarding barriers and facilitators to implementation as determined by participant semi-structured interviews. Barriers and facilitators will serve as a measure of feasibility in Aim 3.
Perceived impact and recommendations | 12 weeks
  Themes regarding perceived impact and recommendations for improvement as determined by participant semi-structured interviews. Perceived impact and recommendations will serve as a measure of acceptability in Aim 3.

OTHER OUTCOMES:
Change in physical function as measured by the Five Times Sit-to-Stand Test | Baseline, 6 weeks
  Time to complete 5 sit-to-stand cycles. This will be used an objective measure of physical function. Assessed at baseline and 6 weeks in Aim 2.
Change in cognitive function as measured by the telephone Montreal Cognitive Assessment (T-MoCA) | Baseline, 6-8 weeks, 12 weeks
  T-MoCA is a validated tool for screening for cognitive impairment by telephone with a range of 0-22 and higher scores indicating better functioning. This will be used as an objective measure of cognitive function. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Change in behavioral activation as measured by the Behavioral Activation for Depression Scale - Short Form (BADS-SF) | Baseline, 6 weeks
  BADS-SF is a validated 9-item self-report measure of behavioral activation. Assessed at baseline and 6 weeks in Aim 2.
Change in engagement in physical, cognitive, and social activities as measured by the Community Healthy Activities Model Program for Seniors questionnaire (CHAMPS) | Baseline, 6-8 weeks, 12 weeks
  CHAMPS is a validated, 40-item scale assesses self-reported physical activity in older adults. The investigators will divide items into physical, cognitive, and social activity to assess engagement across the three target domains of the ACTIVaTE intervention. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Change in quality of life as measured by the CDC Health-Related Quality of Life measure (HRQOL-4) | Baseline, 6 weeks
  4-item validated measure of health-related quality of life. Assessed at baseline and 6 weeks in Aim 2.
Change in depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) | Baseline, 6-8 weeks, 12 weeks
  This 9-item questionnaire is a validated self-report measure of depressive symptoms widely used across settings and populations. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Change in values-aligned living as measured by the Valuing Questionnaire | Baseline, 8 weeks, 12 weeks
  Validated 10-item measure of values-aligned living. Assessed at baseline, 8 weeks, and 12 weeks in Aim 3.
Change in social isolation as measured by the PROMIS Social Isolation Scale (Short Form 4a) | Baseline, 6-8 weeks, 12 weeks
  Validated 4-item measure of subjective social isolation. Assessed at baseline and 6 weeks in Aim 2 and baseline, 8 weeks, and 12 weeks in Aim 3.
Change in global functioning as measured by the World Health Organization Disability Assessment Scale (WHODAS 2.0) | Baseline, 8 weeks, 12 weeks
  Validated 12-item measure of functioning and disability. Assessed at baseline, 8 weeks, and 12 weeks in Aim 3.
Change in care engagement as measured by number of health care visits | Baseline, 8 weeks, 12 weeks
  Self report and chart review of number of primary care visits, psychotherapy/mental health visits, physical therapy/occupational therapy visits, geriatrics visits, and physical activity/recreation program visits. Assessed at baseline, 8 weeks, and 12 weeks in Aim 3.

CONTACTS AND LOCATIONS:
Overall Officials: Meaghan A Kennedy, MD MPH, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No